CLINICAL TRIAL: NCT03444246
Title: A Parallel, Double-blind, Randomized Controlled Trial for the Evaluation of the Treatment and Outcome of Hyperthyroidism With Iodized Salt and Non Iodized Salt
Brief Title: A Trial for the Evaluation of the Treatment and Outcome of Hyperthyroidism With Iodized Salt and Non Iodized Salt
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KY20172032-1
Record Dates: First submitted 2018-02-06; First posted 2018-02-23 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2017-12

CONDITIONS: Hyperthyroidism
MeSH Terms: conditions — Hyperthyroidism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iodine free diet group (Experimental): The arm with non iodized salt，the subject in the non iodized salt group used the iodized salt for the first three months, and the iodized salt was changed after three months.
  Interventions: Dietary Supplement: Iodine free diet group; Dietary Supplement: Normal iodine diet group
- Normal iodine diet group (Active Comparator): The arm with iodized salt，the subject in the control group were consumed with iodized salt within six months.
  Interventions: Dietary Supplement: Normal iodine diet group

INTERVENTIONS:
Dietary Supplement: Iodine free diet group — 120 patients with hyperthyroidism relapsed after new diagnosis or treatment were enrolled. They were randomly divided into iodine free diet group and normal iodine diet group. The two groups were treated with routine antithyroid drugs, followed up for 6 months.
  Arms: Iodine free diet group
Dietary Supplement: Normal iodine diet group — 120 patients with hyperthyroidism relapsed after new diagnosis or treatment were enrolled. They were randomly divided into iodine free diet group and normal iodine diet group. The two groups were treated with routine antithyroid drugs, followed up for 6 months.

SUMMARY:
To clarify the influence of iodine intake in salt on the incidence and treatment of hyperthyroidism patients, so as to provide theoretical basis for accurate formulation of iodine intake in salt, and provide strategies for effective prevention and control of hyperthyroidism.

ELIGIBILITY:
Inclusion Criteria:

1. sign informed consent before any research procedure is carried out
2. men or women aged 18-65 (equal) at the age of 1.
3. had been diagnosed as Graves hyperthyroidism
4. patients with hyperthyroidism who had not been treated with drugs or stopped taking medicine for more than 3 months
5. reduction to the current dose of hyperthyroidism for more than 2 months

Exclusion Criteria:

1. during the period of pregnancy and lactation, those who plan to be pregnant during the study are not granted medical permission.

   Effective contraceptives
2. for the last 1 months or the need for long-term use of amiodarone
3. the history of anaphylaxis (such as systemic anaphylaxis, vasoedema, epidermal exfoliation) Etc.)
4. consecutive use of beta receptor blockers for the last 2 weeks
5. over the past six months, systemic use of corticosteroids (oral or intravenous) is continuous More than 7 days
6. there was an obvious liver disease, showing one of the following cases: two consecutive weeks before A. visits.

It was confirmed that the measurements of AST or ALT were more than 3 times higher than the highest normal value (local data).

B. bilirubin synthesis and / or excretion disorders (such as hyperbilirubinemia), and other Decompensated liver diseases such as coagulation disorders, hepatic encephalopathy, hypoproteinemia, ascites, and esophagus Bleeding from varicose veins. C. acute viral, active, alcoholic, and alcoholic Other types of hepatitis 7 visits for 4 weeks before the 1 (or the local data), leukopenia (less than 3 * 10 9 /L) B/ 0 edition of the First Affiliated Hospital of The Fourth Military Medical University The First Affiliated Hospital, the Fourth Military Medical University B/0 Edition Seventh pages / 13 Pages Or neutropenia (less than 1.5 * 10 9 /L) 8 congestive heart failure at grade III or IV of the New York Heart Association (NYHA) 9 the past 3 months of visit to 1 had a major cardiovascular history, defined as: myocardial infarction Plug and coronary angioplasty or bypass surgery, valvular disease or repair, instability Angina pectoris, transient ischemic attack, or cerebrovascular accident 10 non well controlled atrial fibrillation 11 diagnosis of malignant tumors over the past 5 years 12 history of medullary thyroid carcinoma 13 organ transplantation or AIDS history 14 severe exophthalmos has influenced visual acuity 15 over the last 12 months, there is a history of alcohol abuse or drug abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-03-01 (Estimated); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
Compare the recurrence rate of hyperthyroidism in the two groups | The recurrence rate of hyperthyroidism in the two groups was compared after the first six months of the trial.
  The patients were randomly divided into the non-iodine diet group, the normal iodine diet group, and the two groups were given routine anti-thyroid medication for 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Fourth Military Medical university, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided